CLINICAL TRIAL: NCT01349140
Title: EXPAREL Dose-Response for Single-Injection Femoral Nerve Blocks: A Pharmacodynamics Investigation in Healthy Volunteers
Brief Title: EXPAREL Dose-Response for Single-Injection Femoral Nerve Blocks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EXPAREL Dose-Response
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Each subject is assigned two possible doses between 0-80 mg by the investigators based on previous participants' responses to various doses; and, the dominant side is then randomized to either the higher or lower dose. The response for each dose is the primary interest, and not a comparison of the left vs. the right or different dose combinations within each subject. In other words, of interest are the different doses effects on muscle strength and skin sensitivity across participants (eg., Dose A vs Dose B vs Dose C, etc).
Masking Description: Investigational Drug Service prepared all study medication, with each dose provided to the caregivers in a 30-mL syringe with IV line extension tubing, both wrapped in opaque tape to retain masking since the relative study drug concentration could be inferred by the opacity of the injectate. One syringe was labeled "Dominant" and the other labeled "Other." In this manner, all investigators, nursing staff, and subjects remained masked to the specific concentration/dose during all outcome measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nerve Block (Experimental): The dominant side (left or right) will be randomized to one of two treatment groups: the higher or lower concentration of the local anesthetic EXPAREL. The non-dominant contralateral side will receive the other possible treatment. The volume of each and every single-injection femoral nerve block will be 30 mL (standard for femoral nerve blocks is 30-40 mL).3 Since volume will remain constant, we will vary the dose of EXPAREL by varying concentration (volume x concentration = dose). Of note, EXPAREL may be mixed with normal saline to vary the concentration. Randomization will be based on computer-generated codes. Randomization will be in blocks of two, and stratified by sex.
  Interventions: Drug: SKY0402

INTERVENTIONS:
Drug: SKY0402 — Single-injection femoral nerve block. Initial doses of SKY0402 will begin at 0 mg, and 2 mg (high) for the first subject; and 1 mg (low) and 3 mg (high) for the second subject. The next doses will be between 0-80 mg per side, determined prior to randomization of each subsequent subject. The specific subsequent doses will increase, remain the same, or decrease, determined by the P.I. in consultation with the manufacturer of SKY0402. Doses will always remain within the range of 0-80 mg per side, for a total possible dose of 0-160 mg.
  Other Names: EXPAREL

SUMMARY:
EXPAREL™, an investigational drug product, is a new formulation of a local anesthetic (numbing medicine) that is designed to be longer acting than the currently-available local anesthetics. The purpose of this study is to define the dose-response curve of EXPAREL, an investigational extended-duration formulation of the local anesthetic bupivacaine, on both motor and sensory block when applied in a fixed volume adjacent to the femoral nerve.

DETAILED DESCRIPTION:
Putting local anesthetic next to a nerve is a common way of decreasing the pain that patients feel after surgery. For knee surgery, the local anesthetic is placed next to the femoral nerve in the middle of the crease where the leg meets the body when bending at the hip joint. However, the local anesthetic takes away not only sensation-and therefore pain-but also motor control, leaving muscles weaker. It would greatly improve patient safety if the investigators could administer a very long-acting local anesthetic that decreased postoperative pain, but affected muscle strength only minimally. The purpose of this study is to define the dose-response curve of EXPAREL (also termed SKY0402), an investigational extended-duration formulation of the local anesthetic bupivacaine, on both motor and sensory block when applied in a fixed volume adjacent to the femoral nerve.

This investigation will be a Phase 1, prospective, double-masked, human-subjects dose-response clinical trial.

Enrollment. Subjects will be volunteers of both sexes, age 18 and older. If a volunteer meets inclusion/exclusion criteria and desires study participation, written, informed consent will be obtained. Selection for inclusion will not be based on race or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status.

Subject preparation. Following written, informed consent, subjects will be admitted to the UCSD CTRI and have demographic/morphometric data recorded (e.g., age, weight, height), a medical history recorded, and a brief physical examination. Block placement itself may occur either in the UCSD CTRI or Hillcrest Outpatient Surgical Center Post Anesthesia Care Unit (PACU: this is where regional anesthetics are administered on a regular basis for surgical patients). If the blocks are placed in the PACU, subjects will remain there for two hours and then moved (accompanied by a physician) on their gurney to the UCSD CTRI where they will spend the remainder of the study period. Women of childbearing potential will have a urine pregnancy test. Prior to dosing, baseline quadriceps strength and sensory level measurements will also be obtained. An intravenous line will be placed in an upper extremity, followed by external monitors (pulse oximeter, blood pressure, and EKG), and oxygen by nasal cannula (1-6 L/min). Sedation will be provided by a combination of one or more of the following, titrated to effect: oral valium (10 mg), intravenous fentanyl (50 mcg), and/or intravenous midazolam (1 mg). Following sterile preparation with chlorhexidine gluconate and isopropyl alcohol, and once the topical antiseptic is dry, subjects will have bilateral, single-injection, ultrasound-guided femoral nerve blocks placed using standard UC San Diego techniques as previously published by the current P.I.

Treatment Group Assignment. The dominant side (left or right) will be randomized to one of two treatment groups: the higher or lower concentration of the local anesthetic SKY0402. The non-dominant contralateral side will receive the other possible treatment. The volume of each and every single-injection femoral nerve block will be 30 mL (standard for femoral nerve blocks is 30-40 mL). Since volume will remain constant, we will vary the dose of SKY0402 by varying concentration (volume x concentration = dose). Of note, SKY0402 may be mixed with normal saline to vary the concentration. Randomization will be based on computer-generated codes. Randomization will be in blocks of two.

Dose Determination. Initial doses of SKY0402 will begin at 0 mg (low: exclusively normal saline as the treatment) and 2 mg (high) for the first subject; and 1 mg (low) and 3 mg (high) for the second subject. Since the volume of each of the bilateral blocks will be 30 mL, the first subject's concentrations will be 0 mg / 30 mL (0%) and 2 mg / 30 mL (0.007%); while the second subject's concentrations will be 1 mg / 30 mL (0.003%) and 3 mg / 30 mL (0.010%). Unmasking of treatments will occur following data collection for each subject to allow determination of dosing for subsequent subjects. The subsequent doses will be between 0-160 mg (0.534%) per side, determined prior to randomization of each subsequent subject. The specific subsequent doses will increase, remain the same, or decrease, determined by the P.I. in consultation with the manufacturer of SKY0402. Since the dose-response for SKY0402 remains unknown for single-injection peripheral nerve blocks, a set "tier" or dose-increase plan prior to experience with each subject is impossible. However, the dose will never be increased by more than 20 mg for each side. In addition, doses will always remain within the range of 0-160 mg (0% - 0.534%) per side, and never exceed a total dose of 160 mg for both sides combined. Dose escalation will be stopped and only lower doses will be administered subsequently, if either of the following occurs after study drug administration: one subject experiences clinically significant motor block persisting more than 7 days or four consecutive subjects experience clinically significant motor block persisting more than 5 days.

For unsuccessful local anesthetic deposition (defined as local anesthetic that could not be deposited immediately adjacent to the femoral nerve as viewed by real-time ultrasound) or subject withdrawal from the study, the subjects' data will not be included in the analysis and the subject dropped from the study (subjects will always receive compensation for at least one night in the CTRI--$400-even if they are discharged the day of block placement due to failed deposition). Remaining subjects will remain within the CTRI and within their bed until discharged home. Discharge will occur when quadriceps strength has returned to at least 80% of its baseline value. We consider a difference of less than 20 percentage points to be clinically relevant because a 10% side-to-side strength difference is common, yet functionally unnoticeable in healthy individuals.4,5 Discharge will occur-at the very earliest-24 hours following initial block placement. Therefore, the amount of time subjects will spend in the CTRI will depend upon the duration of local anesthetic action, which will be variable among subjects and is currently unpredictable without a dose-response curve for peripheral nerve blocks using SKY0402. We anticipate the duration of study participation for each subject to be approximately 72 hours. Subjects may withdraw from participation at any time, and will receive compensation for the time they have participated up until withdrawal (subjects who withdraw the day of block placement will receive $400). However, if the research coordinator who is responsible for distributing the compensation is not available at the time of study withdrawal, then the subject will need to return to the CTRI the following day (or following Monday if withdrawal occurs over the weekend) for compensation.

Outcome Measurements. We have selected measures that have established reliability and validity. Staff blinded to treatment group assignment will perform all measures and assessments. For all measurements, the dominant side will always be tested first, followed by the contralateral side. Measurements will be performed prior to local anesthetic administration initiation ("baseline"; Hour 0); as well as specific post-block time points:

Hour Prior to Hour 0 0 0:10 0:20 0:30 0:40 0:50

1 1:15 1:30 1:45 2 2:30 3 3:30 4 5 6 7 8 9 10 24 (Day #2) 27-36 48 (Day #3) 51-60 72 (Day #4) 75-84 96 (Day #5) 99-108 120 (Day #6)

Primary Outcome Measurement

Quadriceps femoris muscle strength: Evaluated using a portable isometric force dynamometer to measure the maximum voluntary isometric contraction (MVIC) in a seated position with the knee flexed at 90º. This variable will be presented and analyzed as post / pre x 100. For all measurements, subjects will be asked to take 2 sec to come to maximum effort contracting the target muscle(s), maintain this effort for 5 sec, and then relax.

Secondary Outcome Measurement

Sensory level: Evaluated using transcutaneous electrical stimulation (TES) in the same manner as described throughout the anesthesia literature (this is a "gold standard" for regional anesthesia studies). After clipping any hair, EKG pads will be positioned 2 cm medial to the proximal patella and quadriceps tendon and attached to a nerve stimulator. The current will be increased from 0 mA until the subject identifies slight discomfort, at which time the current is recorded as the TES value and the nerve stimulator turned off. The secondary end point will be the post-administration maximum current (absolute values in mA).

Safety Assessments Safety assessments will include monitoring of AEs, SAEs, and vital signs (heart rate, respiratory rate, and blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years old
* able and willing to have bilateral femoral nerve blocks placed and repeated motor/sensory testing for 24-120 hours (1-5 days), requiring 1-5 overnight stay(s) in the UCSD CTRI to allow dissipation of local anesthetic infusion effects to near-baseline values
* have the ability to adequately communicate with all study personnel
* willing and capable of providing written informed consent

Exclusion Criteria:

* daily analgesic use for over one week within the past 6 months
* opioid use within the previous 4 weeks
* any neuro-muscular deficit of either femoral nerves and/or quadriceps muscles
* body mass index > 30 kg/m2
* current pregnancy
* incarceration
* any coagulation disorder
* uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigators, may interfere with study assessments or adherence
* any previous allergic reaction to fentanyl, midazolam, or an amide local anesthetic (bupivacaine is of the amide local anesthetic class)
* any previous participation in a SKY0402/EXPAREL study
* nursing mothers
* suspected or known drug or alcohol abuse within the previous year; and/or
* planning on becoming pregnant in the one month following study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University California San Diego
Locations (1):
- UCSD Medical Center Hillcrest, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilfeld BM, Eisenach JC, Gabriel RA. Clinical Effectiveness of Liposomal Bupivacaine Administered by Infiltration or Peripheral Nerve Block to Treat Postoperative Pain. Anesthesiology. 2021 Feb 1;134(2):283-344. doi: 10.1097/ALN.0000000000003630. PMID 33372949
- [Background] Ilfeld BM, Gabriel RA, Eisenach JC. Liposomal Bupivacaine Infiltration for Knee Arthroplasty: Significant Analgesic Benefits or Just a Bunch of Fat? Anesthesiology. 2018 Oct;129(4):623-626. doi: 10.1097/ALN.0000000000002386. No abstract available. PMID 30102616
- [Result] Ilfeld BM, Malhotra N, Furnish TJ, Donohue MC, Madison SJ. Liposomal bupivacaine as a single-injection peripheral nerve block: a dose-response study. Anesth Analg. 2013 Nov;117(5):1248-56. doi: 10.1213/ANE.0b013e31829cc6ae. PMID 24108252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled 14 subjects, and therefore "Protocol Enrollment" is "14". However, each leg of each subject was treated separately with a different dose of liposomal bupivacaine (Exparel); and, therefore the number of units analyzed is 28.
Units Other Than Participants: Side (left or right)
Groups:
- Nerve Block: EXPAREL: active liposome bupivacaine
Period: Overall Study
Arm/Group | Nerve Block
Started | 14; 28 Side (left or right) (We enrolled 14 subjects, and therefore "Protocol Enrollment" is "14". However, each leg of each subject was treated separately with a different dose of liposomal bupivacaine (Exparel); and, therefore the number of units for each subject was 2 and the total number of units analyzed was 28.)
Completed | 14; 28 Side (left or right) (We enrolled 14 subjects, and therefore "Protocol Enrollment" is "14". However, each leg of each subject was treated separately with a different dose of liposomal bupivacaine (Exparel); and, therefore the number of units for each subject was 2 and the total number of units analyzed was 28.)
Not Completed | 0; 0 Side (left or right)

BASELINE CHARACTERISTICS:
Groups:
- Nerve Block: Exparel: liposome bupivacaine
Arm/Group | Nerve Block
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 35 [20 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Femoris Muscle Strength
Description: A dynamometer was used to measure the force produced during a maximum voluntary isometric contraction (MVIC) in a seated position with the knees flexed at 90°. The dynamometer was placed on the anterior tibia perpendicular to the tibial crest, just proximal to the medial malleolus. Subjects were asked to take 2 seconds to come to maximum effort contracting the ipsilateral quadriceps femoris, maintain this effort for 5 seconds, and then relax. The measurements immediately before study drug administration were designated baseline, and all subsequent are expressed as a percentage of the baseline.
Time Frame: Baseline until 99 hours
Population: Each of 14 subjects had a different dose of medication administered to each the left and right sides, and therefore there were 14 subjects, 28 units analyzed.
Measure: Number; unit: percentage of baseline measurement
Units Other Than Participants: side of the body (left or right)
Arm/Group | Nerve Block
Number analyzed (Participants) | 14
Number analyzed (side of the body (left or right)) | 28
percentage of baseline measurement
  Leg #1: Dose 0 mg nondominant | NA — Unavailable due to observation error by research nurse.
  Leg #2: Dose 0 mg nondominant | NA — Unavailable due to observation error by research nurse.
  Leg #3: Dose 0 mg nondominant | 9
  Leg #4: Dose 0 mg dominant | 13
  Leg #5: Dose 1 mg dominant | 12
  Leg #6: Dose 2 mg Nondominant | NA — Unavailable due to observation error by research nurse.
  Leg #7: Dose 3 mg Dominant | 8
  Leg #8: Dose 4 mg dominant | NA — Unavailable due to observation error by research nurse.
  Leg #9: Dose 7 mg nondominant | NA — Unavailable due to observation error by research nurse.
  Leg #10: Dose 10 mg nondominant | NA — Unavailable due to observation error by research nurse.
  Leg #11: Dose 15 mg dominant | NA — Unavailable due to observation error by research nurse.
  Leg #12: Dose 20 mg dominant | NA — Unavailable due to observation error by research nurse.
  Leg #13: Dose 25 mg dominant | 31
  Leg #14: Dose 30 mg dominant | 52
  Leg #15: Dose 35 mg nondominant | 27
  Leg #16: Dose 40 mg nondominant | 74
  Leg #17: Dose 40 mg nondominant | 49
  Leg #18: Dose 50 mg nondominant | 13
  Leg #19: Dose 60 mg dominant | 52
  Leg #20: Dose 60 mg dominant | 28
  Leg #21: Dose 60 mg dominant | 39
  Leg #22: Dose 60 mg nondominant | 60
  Leg #23: Dose 70 mg dominant | 40
  Leg #24: Dose 80 mg dominant | 9
  Leg #25: Dose 80 mg dominant | 81
  Leg #26: Dose 80 mg nondominant | 41
  Leg #27: Dose 80 mg nondominant | 11
  Leg #28: Dose 80 mg nondominant | 37

2. Secondary Outcome: Sensory Effect
Description: We evaluated tolerance of transcutaneous electrical stimulation with the same quantitative procedure as described previously. Electrocardiogram pads were placed 2 cm medial to the distal quadriceps tendon and attached to a nerve stimulator (EZstimII, Model ES400; Life-Tech, Stafford, TX). The current was increased from 0 mA until subjects described mild discomfort, at which time the current was recorded as the tolerated level and the nerve stimulator turned off. All sensory measurements are expressed as a percentage of each patient's pre-infusion baseline.
Time Frame: Baseline until 99 hours
Population: as for outcome 1
Measure: Number; unit: percentage of baseline measurement
Units Other Than Participants: side of the body (left or right)
Arm/Group | Nerve Block
Number analyzed (Participants) | 14
Number analyzed (side of the body (left or right)) | 28
percentage of baseline measurement
  Leg #1: Dose 0 mg nondominant | 127
  Leg #2: Dose 0 mg nondominant | 275
  Leg #3: Dose 0 mg nondominant | 486
  Leg #4: Dose 0 mg dominant | 209
  Leg #5: Dose 1 mg dominant | 400
  Leg #6: Dose 2 mg Nondominant | NA — Subject never exhibited a sensory block >100% of baseline
  Leg #7: Dose 3 mg Dominant | NA — Subject never exhibited a sensory block >100% of baseline
  Leg #8: Dose 4 mg dominant | 125
  Leg #9: Dose 7 mg nondominant | NA — Subject never exhibited a sensory block >100% of baseline
  Leg #10: Dose 10 mg nondominant | 127
  Leg #11: Dose 15 mg dominant | 300
  Leg #12: Dose 20 mg dominant | 156
  Leg #13: Dose 25 mg dominant | 107
  Leg #14: Dose 30 mg dominant | NA — Subject never exhibited a sensory block >100% of baseline
  Leg #15: Dose 35 mg nondominant | 225
  Leg #16: Dose 40 mg nondominant | NA — Subject never exhibited a sensory block >100% of baseline
  Leg #17: Dose 40 mg nondominant | 109
  Leg #18: Dose 50 mg nondominant | 300
  Leg #19: Dose 60 mg dominant | 150
  Leg #20: Dose 60 mg dominant | 190
  Leg #21: Dose 60 mg dominant | 157
  Leg #22: Dose 60 mg nondominant | 200
  Leg #23: Dose 70 mg dominant | 229
  Leg #24: Dose 80 mg dominant | 363
  Leg #25: Dose 80 mg dominant | 325
  Leg #26: Dose 80 mg nondominant | 150
  Leg #27: Dose 80 mg nondominant | 200
  Leg #28: Dose 80 mg nondominant | 138

ADVERSE EVENTS:
Arm/Group | Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nerve Block (N=14)
rash (Skin and subcutaneous tissue disorders) | 1 (1) — rash in participant who received saline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No